CLINICAL TRIAL: NCT03752177
Title: A Phase 1a/1b Study of LY3415244, a Bispecific Antibody in Patients With Advanced Solid Tumors
Brief Title: A Study of LY3415244 in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated during dose escalation after a determination was made that the risk:benefit ratio no longer favored continued evaluation.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17099; J1C-MC-JZDA (Other: Eli Lilly and Company); 2018-001598-25 (EudraCT Number)
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Results first posted 2021-08-31 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Solid Tumor
Keywords: TIM-3; PD-L1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3415244 Dose Escalation (Experimental): Participants received 3 milligrams (mg) LY3415244 (Cohort A1), 10 mg LY3415244 (Cohort A2), 30 mg LY3415244 (Cohort A3) and 70 mg LY3415244 (Cohort A4) as an intravenous (IV) infusion on day (D)1 and D15 of each 28-day cycle every 2 weeks (Q2W).
  Interventions: Drug: LY3415244
- LY3415244 Dose Expansion (Experimental): Phase 1b dose expansion was planned but not initiated as dose escalation ended at cohort A4. Study did not achieve its primary objective of establishing a recommended phase 2 dose (RP2D) due to early termination of the study by Cohort A4.
  Interventions: Drug: LY3415244

INTERVENTIONS:
Drug: LY3415244 — Administered IV

SUMMARY:
The goal of this study is to evaluate the safety of LY3415244, a PD-L1/TIM-3 bispecific antibody, administered as monotherapy to participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* For Phase 1a/b, histologic or cytologic confirmation of advanced solid tumor.
* For Phase 1a/b, biopsy of tumor samples are required. Newly obtained core or excisional biopsy of a tumor lesion prior to study enrollment and undergo a biopsy procedure during the study.
* Phase 1a, prior anti-PD-1 or anti-PD-L1 therapy or other immunotherapy is allowed.
* Phase 1b, prior anti-PD-1 or anti-PD-L1 therapy is required where anti-PD-1 or anti-PD-L1 is standard of care in respective tumor types if the following criteria are met:

  * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy
  * Must have completely recovered to baseline level prior to screening from any adverse events (AEs) that occurred from receiving prior immunotherapy
  * Must not have experienced a Grade ≥3 immune-related AE or immune related neurologic or ocular AE, pneumonitis or cardiomyopathy of any grade while receiving prior immunotherapy
  * Must not have required immunosuppressive agent, other than corticosteroids for the management of an adverse event and not currently require maintenance doses of >10 milligrams (mg) prednisone (or equivalent) per day
* Must have at least 1 measurable lesion as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Have adequate organ function.
* Have an estimated life expectancy ≥12 weeks, in the judgement of the investigator.

Exclusion Criteria:

* Have symptomatic central nervous system (CNS) malignancy or metastasis not requiring concurrent treatment, including but not limited to surgery, radiation, corticosteroids and/or anticonvulsants to treat CNS metastases, and their disease is asymptomatic and radiographically stable for at least 30 days.
* Have received a live vaccine within 30 days before the first dose of study treatment.
* If female, is pregnant, breastfeeding, or planning to become pregnant.
* Have a history or current evidence of any condition, therapy, or laboratory abnormality that might interfere with the participant's participation.
* Have moderate or severe cardiovascular disease.
* Have a serious concomitant systemic disorder that would compromise the participant's ability to adhere to the protocol, including known infection with human immunodeficiency virus (HIV), active hepatitis B virus (HBV), active hepatitis C virus (HCV), active autoimmune disorders, or prior documented severe autoimmune or inflammatory disorders requiring immunosuppressive treatment.
* Use of escalating or chronic supraphysiologic doses of corticosteroids or immunosuppressive agents (such as, cyclosporine). [Use of topical, ophthalmic, inhaled, and intranasal corticosteroids permitted].
* Bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection.
* Evidence of interstitial lung disease or noninfectious pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chuo-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3415244 in Participants With Advanced Solid Tumors — https://www.lillytrialguide.com/en-US/studies/solid-tumor/JZDA

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 1a of study consisted of dose-escalation assessment and Phase 1b of study included dose expansion. Four out of planned eight cohorts (one optional) in Phase 1a were completed. Phase 1b dose expansion was planned but not initiated as dose escalation ended at cohort A4.A participant completed study if they completed at least 1 cycle (28 days).
Groups:
- Cohort A1: Participants received 3 milligrams (mg) LY3415244 as an intravenous (IV) infusion on day (D)1 and D15 of each 28-day cycle every 2 weeks (Q2W).
- Cohort A2: Participants received 10 mg LY3415244 as an IV infusion on D1 and D15 of each 28-day cycle Q2W.
- Cohort A3: Participants received 30 mg LY3415244 as an IV infusion on D1 and D15 of each 28-day cycle Q2W.
- Cohort A4: Participants received 70 mg LY3415244 as an IV infusion on D1 and D15 of each 28-day cycle Q2W.
Period: Overall Study
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4
Started | 3 | 3 | 3 | 3
Received at Least 1 Dose of Study Drug | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.33 (2.31) | 57.00 (11.36) | 48.33 (20.60) | 55.67 (3.79) | 53.58 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 1 | 6
  Male | 1 | 1 | 2 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 3 | 1 | 8
  Unknown or Not Reported | 1 | 1 | 0 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 2 | 3 | 2 | 8
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 1 | 2 | 2 | 5
  United States | 1 | 1 | 1 | 0 | 3
  Japan | 2 | 1 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase1a: Number of Participants With LY3415244 Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as an adverse event (AE) occurring during Cycle 1(28 days) that was considered at least possibly related to study drug, was considered dose-dependent, and fulfilled a criteria selected (using the National Cancer Institute Common Terminology Criteria for Adverse Events,version 4.0 [NCI-CTCAE v 4.0] [NCI 2009]):Grade 3 thrombocytopenia requiring platelet transfusion or grade 4 thrombocytopenia. Grade greater than or equal to (≥) 3 febrile neutropenia, anemia requiring a blood transfusion and any other Grade 4 hematologic toxicity that last >7 days. Grade ≥ 3 colitis or noninfectious pneumonitis, Grade ≥ 3 fatigue lasting >7 days, Grade ≥ 3 hypertension despite of maximal medical therapy. Grade 4 immune-related adverse event (irAE), liver transaminase elevation >8x upper limit of normal (ULN) or total bilirubin >3x ULN.
Time Frame: Baseline through Cycle 1 (28 Day Cycle)
Population: All participants who received at least 1 dose of study drug and had evaluable DLT data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4
Number analyzed (Participants) | 3 | 3 | 3 | 2
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Phase1a: Pharmacokinetics (PK): Minimum Concentration (Cmin) of LY3415244
Description: Cmin of LY3415244 was evaluated.
Time Frame: Cycle 1 Day 1 (C1D1) and C1D15: pre-dose, 2 hours(h), 4h, 24h, 72h, 120h and 168h post-dose; C2D1, C2D15, C3D1, C3D15, C4D1, C4D15, C5D1, C5D15, C6D1 and C6D15: pre-dose
Population: All participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4
Number analyzed (Participants) | 3 | 3 | 3 | 3
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 3
  Cycle 1 Day 1 |  |  | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual value of Cmin = 5790 ng/mL. | 4270 (26)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 1 | 2 | 0
  Cycle 1 Day 15 |  | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual value of Cmin = 151 ng/mL. | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of Cmin = 146 ng/mL, 8240 ng/mL. |

3. Secondary Outcome: Phase1b: Objective Response Rate (ORR): Percentage of Participants Who Achieve Complete Response (CR) or Partial Response (PR)
Description: ORR was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline through Measured Progressive Disease (Up To 24 Months)
Population: Zero participants were analyzed for this outcome. Data were not captured as study was terminated early and no participant were enrolled into Phase 1b expansion.
Arm/Group | LY3415244 Dose Expansion
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase1b: Duration of Response (DoR)
Description: Duration of response was defined using RECIST v. 1.1 criteria as the time from the date criteria were met for the first objectively recorded CR or PR until the first date criteria for PD were met or death from any cause. CR was the disappearance of all lesions and pathological lymph node reduction in the short axis to <10 mm. PR was a ≥30% decrease in the sum of the diameters of target lesions. PD was a ≥20% increase in the sum of the diameters of target lesions with the sum demonstrating an absolute increase of ≥5 mm; the appearance of ≥1 new lesions or unequivocal progression of non-target lesions. Participants who were not known to have died and who did not have PD were censored at the date of the last tumor assessment prior to the date of any subsequent systemic anticancer therapy.
Time Frame: Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Up To 24 Months)
Population: as for outcome 3
Arm/Group | LY3415244 Dose Expansion
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase1b: Time to Response (TTR)
Description: Data were not captured as study was terminated early and no participant were enrolled into Phase 1b expansion. Time to treatment response was defined as date of first dose of study drug to the date of confirmed complete response (CR) or partial response (PR) using Response evaluation Criteria in Solid Tumors (RECIST v1.0) criteria. CR was defined as the disappearance of all target and non-target lesions and normalization of tumor marker levels in non-target lesions. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Baseline to Date of CR or PR (Up To 24 Months)
Population: as for outcome 3
Arm/Group | LY3415244 Dose Expansion
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase1b: Disease Control Rate (DCR): Percentage of Participants With a Best Overall Response of CR, PR, and Stable Disease
Description: DCR is the percentage of participants with a best overall response of CR, PR or stable disease (SD) as defined by RECIST v1.1. CR is defined as disappearance of all target and non-target lesions and no appearance of new lesions.PR is defined as at least a 30% decrease in sum of longest diameter (LD) of target lesions (taking as reference the baseline sum LD),no progression of non-target lesions, and no appearance of new lesions.SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm,or unequivocal progression of non-target lesions,or 1 or more new lesions.
Time Frame: Baseline through Measured Progressive Disease (Up To 24 Months)
Population: as for outcome 3
Arm/Group | LY3415244 Dose Expansion
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase1b: Progression Free Survival (PFS)
Description: Progression-free survival time was measured from treatment start until the date of objective progression as defined by Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1), or death from any cause. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. Patients who have neither progressed nor died were censored at the day of their last radiographic tumor assessment, if available, or date of treatment start if no post-baseline radiographic assessment is available.
Time Frame: Baseline to Objective Progression or Death Due to Any Cause (Up To 24 Months)
Population: as for outcome 3
Arm/Group | LY3415244 Dose Expansion
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up To 24 Months
Description: All enrolled participants. Gastrointestinal stoma complication was not treatment related adverse event and the Infusion related reaction is treatment related adverse event.
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4
All-Cause Mortality (participants affected / at risk) | 2/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1 (N=3) | Cohort A2 (N=3) | Cohort A3 (N=3) | Cohort A4 (N=3)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1 (N=3) | Cohort A2 (N=3) | Cohort A3 (N=3) | Cohort A4 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye movement disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Phase 1b dose expansion was planned but not initiated as dose escalation ended at cohort A4. Study did not achieve its primary objective of establishing a recommended phase 2 dose (RP2D) due to early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must delay publications until a multi-center publication is disclosed, (or for a time period if no multi-center publication is disclosed).

DOCUMENTS (2):
  • Study Protocol (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT03752177/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT03752177/SAP_001.pdf